CLINICAL TRIAL: NCT00483028
Title: A Randomized Double-Blind, Parallel, Placebo-Controlled Trial to Examine the Efficacy of Oral Donepezil (5 mg QD for 6 Weeks) After Single Dose and Steady State Therapy (2 Weeks and 6 Weeks) in Subjects With Mild Cognitive Impairment
Brief Title: A Randomized, Placebo-Controlled Trial to Examine the Efficacy of Oral Donepezil in Subjects With MCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A9001134
Record Dates: First submitted 2007-06-05; First posted 2007-06-06 (Estimated); Last update posted 2008-02-05 (Estimated); Status verified 2008-02

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

INTERVENTIONS:
Drug: donezepil (Aricept)

SUMMARY:
To purpose of this study is to estimate the effect of donepezil on Neuropsychological Testing (NPT) and brain Proton Magnetic Resonance Spectroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females ages 55-90 inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and heart rate measurement, 12-lead ECG and clinical laboratory tests)
* Body Mass Index (BMI) between 18 to 34 kg/m2, inclusive; and a total body weight
* Subjects with mild cognitive impairment (MCI) must have a reliable informant who has an average of 10 hours per week or more contact with the subject.
* Memory complaints and memory difficulties, which are verified by an informant
* Mini-mental status exam (MMSE) score of 24-30

Exclusion Criteria:

* Subjects with known hypersensitivity to donepezil hydrochloride or to piperidine derivatives
* Insulin-requiring diabetes or uncontrolled diabetes mellitus
* Subjects with a current diagnosis of depression or other psychiatric illnesses

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38
Dates: Start 2004-06; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Neuropsychologic test scores: GMLT, DSST, Cog State TM including PAL test, RAVLT, ADAS-cog at baseline (pre-dose) 5 and 8 hours after the first dose and 2 and 6 weeks. (Continues in next bullet.)
MRS (Magnetic Resonance Spectroscopy) profile including but not limited to NAA (N-acetyl-aspartate), NAA/Cr (N-acetyl-aspartate/creatinine ratio), MI (Myoinositol) and MI/Cr (Myoinositol/creatinine ratio).

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, New Haven, Connecticut
  - Pfizer Investigational Site, Albany, New York

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9001134&StudyName=A+Randomized%2C+Placebo%2DControlled+Trial+to+Examine+the+Efficacy+of+Oral+Donepezil+in+subjects+with+MCI